CLINICAL TRIAL: NCT00006133
Title: Randomized Study of Oral Contraceptives or Hormone Replacement Therapy in Women With Systemic Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Alabama at Birmingham (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/15327; UAB-SELENA
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Estradiol; Ethinyl Estradiol; Medroxyprogesterone; Norethindrone

INTERVENTIONS:
Drug: estradiol
Drug: ethinyl estradiol
Drug: medroxyprogesterone
Drug: norethindrone

SUMMARY:
OBJECTIVES: I. Determine the effect of oral contraceptives containing low-dose synthetic estrogens and progestins on disease activity in premenopausal women with inactive, stable, or moderate systemic lupus erythematosus (SLE).

II. Determine the effect of hormone replacement therapy with conjugated estrogens and progestins on disease activity in postmenopausal women with inactive, stable, or moderate SLE.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to age/menopausal status (35 and under/premenopausal vs 50 and over/postmenopausal). Both strata are randomized to one of two treatment arms.

Stratum 1 (Premenopausal/Oral contraceptives): Patients receive either oral ethinyl estradiol and norethindrone or placebo daily for 28 days beginning on the Sunday following the first day of the menstrual cycle.

Stratum 2 (Postmenopausal/Hormone replacement therapy): Patients receive either oral estradiol and medroxyprogesterone or placebo on days 1-12 monthly.

Treatment continues in both arms of both strata for a total of 13 courses in the absence of a severe disease flare-up or other complication that would preclude further study participation.

All patients are followed at 1 year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Established systemic lupus erythematosus meeting American College of Rheumatology criteria

Inactive disease Systemic Lupus Erythematosus Activity Index (SLEDAI) score no greater than 4

No increase in score of more than 2 from baseline over the past 3 months

Receiving the equivalent of 5 mg or less of prednisone per day OR Stable/active disease SLEDAI score 5-12

No increase in score of more than 2 from baseline over the past 3 months

Prednisone dose up to 0.5 mg/kg/day for control of underlying disease allowed if stable dose for at least 3 weeks

No concurrent severe disease activity as defined by any of the following:

* Acute renal disease (i.e., rising creatinine levels, cellular sediment, or increasing proteinuria)
* Involvement of 3 or more organ systems requiring more than the equivalent of 0.5 mg/kg/day of prednisone
* Necessity of immediate hospitalization for symptom control

No presence of a high titer IgG, IgM, or IgA antiphospholipid antibodies (aPL) GPL and MPL no more than 40 APL no more than 50

No features of primary antiphospholipid antibody syndrome

--Prior/Concurrent Therapy--

Biologic therapy: Not specified

Chemotherapy: Not specified

Endocrine therapy: See Disease Characteristics

Radiotherapy: Not specified

Surgery: Prior hysterectomy allowed

--Patient Characteristics--

Age: 35 and under for oral contraceptive stratum (premenopausal) 50 and over for hormone replacement therapy stratum (postmenopausal)

Menopausal status:

* Premenopausal for oral contraceptive stratum
* Postmenopausal for hormone replacement therapy stratum
* Follicle-stimulating hormone greater than 40 mIU/mL OR Amenorrhea for 6 months

Performance status: See Disease Characteristics

Hematopoietic: Not specified

Hepatic:

* No hepatic dysfunction
* No tumors of the liver

Renal: See Disease Characteristics

Cardiovascular:

* No uncontrolled high blood pressure requiring frequent change in medication
* Concurrent hypertension controlled with stable medication allowed
* No history of spontaneous superficial or deep venous thrombosis or arterial thrombosis
* No prior myocardial infarction
* Oral contraceptive stratum: No angina No diastolic blood pressure greater than 90 mm Hg or systolic blood pressure greater than 140 mm Hg on 3 separate determinations
* Hormone replacement therapy stratum: No diastolic blood pressure greater than 95 mm Hg or systolic blood pressure greater than 145 mm Hg on 3 separate determinations

Pulmonary: No history of pulmonary embolus

Other:

* Not pregnant
* Oral contraceptive stratum: Negative pregnancy test Fertile patients must use effective barrier contraception
* No prior gynecologic malignancy or breast malignancy
* No undiagnosed vaginal bleeding
* No diabetes (present prior to use of glucocorticoids) requiring oral hypoglycemic medications or insulin
* No congenital hyperlipidemia
* No complicated migraines (i.e., associated with neurological sequelae)

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 970
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Graciela S. Alarcon, Study Chair — University of Alabama at Birmingham
Locations (17):
- United States (17):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - University of California-San Francisco, San Francisco, California
  - Pritzker School of Medicine, Chicago, Illinois
  - Louisiana State University School of Medicine, Shreveport, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Hospital for Joint Diseases, New York, New York
  - Saint Luke's-Roosevelt Hospital Center, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Rheumatology Associates of Long Island, Port Jefferson Station, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas- Houston Medical School, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin